CLINICAL TRIAL: NCT06295809
Title: A Phase 2/3, Adaptive, Randomized, Open-label, Clinical Study to Evaluate Neoadjuvant and Adjuvant Intismeran Autogene (mRNA-4157) in Combination With Pembrolizumab (MK-3475) Versus Standard of Care, and Pembrolizumab Monotherapy in Participants With Resectable Locally Advanced Cutaneous Squamous Cell Carcinoma (LA cSCC) (INTerpath-007)
Brief Title: A Study of (Neo)Adjuvant Intismeran Autogene (V940) and Pembrolizumab in Cutaneous Squamous Cell Carcinoma (V940-007)
Acronym: INTerpath-007
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V940-007; 2023-505712-37-00 (Registry Identifier: EU CT); U1111-1292-3589 (Registry Identifier: UTN); V940 (Other: MSD)
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Squamous Cell; Skin Neoplasms
Keywords: pembrolizumab
MeSH Terms: conditions — Carcinoma, Squamous Cell; Skin Neoplasms | interventions — pembrolizumab; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab plus Intismeran autogene with SOC (Experimental): Participants will receive intismeran autogene 1 mg intramuscular (IM) injection every 3 weeks (q3w) for up to 6 weeks and pembrolizumab 400 mg intravenous (IV) infusion every 6 weeks (q6w) up to 12 weeks as neoadjuvant therapy prior to surgery; followed by intismeran autogene 1 mg IM injection q3w up to 21 weeks.
  Interventions: Biological: Pembrolizumab; Biological: Intismeran autogene; Procedure: Surgery
- Standard of Care (SOC) (Active Comparator): Participants will receive surgical resection as per local guidelines with/without adjuvant radiation therapy (RT) at investigator's discretion.
  Interventions: Procedure: Surgery
- Pembrolizumab with SOC (Experimental): Participants will receive pembrolizumab 400 mg IV infusion q6w up to 12 weeks as neoadjuvant therapy prior to surgery.
  Interventions: Biological: Pembrolizumab; Procedure: Surgery

INTERVENTIONS:
Biological: Pembrolizumab — IV Infusion
  Other Names: MK-3475; Keytruda®
  Arms: Pembrolizumab plus Intismeran autogene with SOC; Pembrolizumab with SOC
Biological: Intismeran autogene — IM injection
  Other Names: mRNA-4157; V940
  Arms: Pembrolizumab plus Intismeran autogene with SOC
Procedure: Surgery — Local resection of cancerous lesions of the skin

SUMMARY:
This is a two-part (Phase 2/Phase 3) study of intismeran autogene, an individualized neoantigen therapy (INT), plus pembrolizumab in participants with locally resectable advanced cutaneous squamous cell carcinoma (LA cSCC). Phase 2 has three arms intismeran autogene plus pembrolizumab given as neoadjuvant and adjuvant treatment with standard of care (SOC), standard of care (surgical resection with/without adjuvant radiation therapy (RT) only at investigator's discretion) and pembrolizumab monotherapy given as neoadjuvant and adjuvant treatment with SOC. This phase will assess the safety and efficacy of intismeran autogene in combination with pembrolizumab as neoadjuvant and adjuvant therapy in participants with resectable LA cSCC as compared to standard of care SOC only. The primary hypothesis is that intismeran autogene plus pembrolizumab with SOC is superior to SOC only with respect to event free survival (EFS) as assessed by the investigator. Phase 3 expansion will be determined by prespecified Go-No-Go decision in which 412 additional participants will be randomized to intismeran autogene plus pembrolizumab with SOC and SOC only, without changing the inclusion/exclusion criteria for the additional enrollment or study endpoints.

As of Amendment 04, enrollment was stopped and there will be no Phase 3 expansion.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed diagnosis of resectable cSCC as the primary site of malignancy (metastatic skin involvement from another primary cancer or from an unknown primary cancer is not permitted).
* Has LA Stage II-IV (M0) cSCC without distant metastases.
* cSCC must be amenable to surgery (resectable) with curative intent.
* Has a formalin-fixed, paraffin-embedded (FFPE) tumor sample available or is able to provide one that is suitable for the Next-generation Sequencing (NGS) required for this study.
* For males, agrees to be abstinent from penile-vaginal intercourse OR agrees to use a highly effective contraceptive method while receiving adjuvant radiation therapy (RT), and for ≥3 months after the last dose of study intervention
* Is female and not pregnant/breastfeeding and at least one of the following applies during the study : is not a woman of childbearing potential (WOCBP), is a WOCBP and uses highly effective contraception (low user dependency method OR a user dependent hormonal method in combination with a barrier method) at least during use of intismeran autogene: 15 days, Pembrolizumab: 120 days, Adjuvant RT, if performed: 90 days after last exposure or is a WOCBP who is abstinent from heterosexual intercourse.
* Has measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology.
* Has a life expectancy of >3 months per investigator assessment.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 14 days before randomization.
* Has adequate organ function.
* If hepatitis B surface antigen (HBsAg) positive, must have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization
* If there is a history of hepatitis C virus (HCV) infection, HCV viral load must be undetectable at screening
* If human immunodeficiency virus (HIV)-infected, must have well controlled HIV on antiretroviral therapy (ART)

Exclusion Criteria:

* Has any other histologic type of skin cancer other than invasive cSCC as well as mixed histology, eg, basal cell carcinoma that has not been definitively treated with surgery or radiation, Bowen's disease, Merkel cell carcinoma (MCC), or melanoma
* Has distant metastatic disease (M1), visceral and/or distant nodal
* Has received prior therapy with an anti-programmed cell death receptor 1 (anti-PD-1), anti-programmed cell death receptor ligand 1 (anti-PD-L1), or anti-programmed cell death receptor ligand 2 (anti-PD-L2) agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte associated protein 4 (CTLA-4), OX-40, CD137)
* Has received prior systemic anticancer therapy including investigational agents for cSCC before randomization
* Has received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 2 weeks of the screening blood sample (including the NGS blood sample)
* Has received prior treatment with another cancer vaccine
* Has received prior radiotherapy to the index lesion (in-field lesion). Must have recovered from all radiation-related toxicities prior to randomization and not have had radiation pneumonitis
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years
* History of chronic lymphocytic leukemia (CLL)
* History of central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to either intismeran autogene or pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid) is allowed
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has HIV with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection
* Has had a myocardial infarction within 6 months of randomization
* History of allogeneic tissue/solid organ transplant
* Has not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | Up to ~22 months
  EFS is defined as the time from randomization to any of the following events as assessed by the investigator: progression of disease that precludes surgery, or inability to undergo R0 or R1 surgical resection; disease recurrence (local, regional, or distant); new primary high-risk cSCC; death due to any cause. EFS will be presented.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to ~22 months
  ORR is defined as the proportion of participants who have a complete response (CR) or partial response (PR). ORR will be presented.
Freedom from surgery (FFS) rate | Up to ~22 months
  FFS rate is defined as the proportion of participants with clinical CR with no residual tumor on clinical exam and imaging with the confirmation of negative biopsy. FFS rate will be presented.
Pathologic complete response (pCR) rate | Up to ~22 months
  pCR rate is defined as the proportion of participants who have complete absence of viable tumor in the surgical resection specimen. The pCR rate will be presented.
Major pathologic response (mPR) rate | Up to ~22 months
  mPR rate is defined as the proportion of participants who have ≤10% of viable tumor cells in the surgical resection specimen. The mPR rate will be presented.
Disease-specific survival (DSS) | Up to ~22 months
  DSS is defined as time from randomization to death due to progression of cancer under study. DSS will be presented.
Overall Survival (OS) | Up to ~22 months
  OS is defined as the time from the date of randomization to death due to any cause. The OS will be reported for all participants.
Percentage of participants who experience an adverse event (AE) | Up to ~22 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Percentage of participants who discontinue study intervention due to AEs | Up to ~22 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue intervention due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (106):
- United States (21):
  - USC/Norris Comprehensive Cancer Center ( Site 1112), Los Angeles, California
  - Hoag Memorial Hospital Presbyterian ( Site 1122), Newport Beach, California
  - Stanford Cancer Center ( Site 1109), Palo Alto, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center ( Site 1103), Sacramento, California
  - Winship Cancer Institute, Emory University ( Site 1151), Atlanta, Georgia
  - University of Iowa-Holden Comprehensive Cancer Center ( Site 1118), Iowa City, Iowa
  - University of Kentucky Chandler Medical Center ( Site 1101), Lexington, Kentucky
  - Ochsner Clinic Foundation ( Site 1113), New Orleans, Louisiana
  - Massachusetts General Hospital ( Site 1162), Boston, Massachusetts
  - Dana-Farber Cancer Institute ( Site 1130), Boston, Massachusetts
  - Washington University School of Medicine-Internal Medicine/Oncology ( Site 1100), St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 1125), Hackensack, New Jersey
  - Atlantic Health System Morristown Medical Center ( Site 1136), Morristown, New Jersey
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 1160), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center ( Site 1121), New York, New York
  - Providence Portland Medical Center ( Site 1102), Portland, Oregon
  - UPMC Hillman Cancer Center ( Site 1107), Pittsburgh, Pennsylvania
  - Avera Cancer Institute- Research ( Site 1161), Sioux Falls, South Dakota
  - University of Virginia Health System ( Site 1115), Charlottesville, Virginia
  - Inova Schar Cancer Institute ( Site 1108), Fairfax, Virginia
  - University Hospital and UW Health Clinics ( Site 1119), Madison, Wisconsin
- Argentina (5):
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 1213), Mar del Plata, Buenos Aires
  - Fundacion Estudios Clinicos-Oncology ( Site 1205), Rosario, Santa Fe Province
  - Sanatorio Finochietto ( Site 1202), Buenos Aires
  - Investigaciones Clinicas Moleculares (ICM) ( Site 1212), CABA
  - Hospital Italiano de Córdoba ( Site 1204), Córdoba
- Australia (7):
  - Melanoma Institute Australia-Clinical Trials Unit ( Site 3205), Wollstonecraft, New South Wales
  - Sunshine Coast University Hospital-Medical Oncology ( Site 3212), Birtinya, Queensland
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Si, Brisbane, Queensland
  - Gold Coast University Hospital-Cancer and Blood Disorders Clinical Trial Team ( Site 3207), Gold Coast, Queensland
  - Gallipoli Medical Research Ltd-GMRF CTU ( Site 3206), Greenslopes, Queensland
  - Austin Health ( Site 3209), Heidelberg, Victoria
  - One Clinical Research ( Site 3211), Nedlands, Western Australia
- Belgium (2):
  - Cliniques universitaires Saint-Luc ( Site 1701), Brussels, Bruxelles-Capitale, Region de
  - UZ Gent-Medical oncology ( Site 1702), Ghent, Oost-Vlaanderen
- Brazil (7):
  - Clinica Amo - Rio Vermelho-INSTITUTO ETICA ( Site 1315), Salvador, Estado de Bahia
  - Hospital de Cancer de Londrina-Clinical Research Unit ( Site 1316), Londrina, Paraná
  - Associação Hospitalar Beneficente São Vicente de Paulo-Instituto do Câncer ( Site 1309), Passo Fundo, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição-Centro Integrado de Pesquisa em Oncologia ( Site 1300), Porto Alegre, Rio Grande do Sul
  - ANIMI - Unidade de Tratamento Oncologico ( Site 1312), Lages, Santa Catarina
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto-Centro Integrado de Pesquisa ( Site, São José do Rio Preto, São Paulo
  - IPITEC ( Site 1313), São Paulo, São Paulo
- Canada (2):
  - Jewish General Hospital ( Site 1009), Montreal, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Univer, Sherbrooke, Quebec
- Chile (4):
  - FALP-UIDO ( Site 1401), Santiago, Region M. de Santiago
  - Clínica Alemana de Santiago-Gynecology and Obstetrics ( Site 1410), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 1411), Temuco, Región de la Araucanía
  - CIDO SpA-Oncology ( Site 1405), Temuco, Región de la Araucanía
- Colombia (3):
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 1501), Medellín, Antioquia
  - Oncologos del Occidente ( Site 1504), Pereira, Risaralda Department
  - Fundación Valle del Lili ( Site 1502), Cali, Valle del Cauca Department
- Vseobecna fakultni nemocnice v Praze-Department of Dermatology ( Site 1800), Prague, Praha 2, Czechia
- France (9):
  - CHU de Bordeaux Hop St ANDRE ( Site 1902), Bordeaux, Aquitaine
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone ( Site 1903), Marseille, Bouches-du-Rhone
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand ( Site 1904), Dijon, Bourgogne-Franche-Comté
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE ( Site 1908), Toulouse, Haute-Garonne
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu-Onco-Dermatology ( Site 1910), Nantes, Loire-Atlantique
  - Hopital Claude Huriez - CHU de Lille ( Site 1907), Lille, Nord
  - centre hospitalier lyon sud ( Site 1901), Pierre-Bénite, Rhone
  - Hôpital Saint-Louis ( Site 1906), Paris
  - Gustave Roussy ( Site 1909), Villejuif, Île-de-France Region
- Germany (8):
  - NCT ( Site 2002), Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen-Hautklinik ( Site 2003), Tübingen, Baden-Wurttemberg
  - klinikum rechts der isar der technischen universität münchen ( Site 2009), München, Bavaria
  - Universitaetsklinikum Wuerzburg-Department of Dermatology ( Site 2001), Würzburg, Bavaria
  - Klinikum Dortmund Klinikzentrum Mitte ( Site 2008), Dortmund, North Rhine-Westphalia
  - Universitaetsklinikum Essen-Klinik für Dermatologie, Venerologie und Allergologie ( Site 2005), Essen, North Rhine-Westphalia
  - Universitätsmedizin Johannes Gutenberg Universität Mainz ( Site 2007), Mainz, Rhineland-Palatinate
  - Universitätsklinikum Schleswig-Holstein-Dermatology ( Site 2012), Lübeck, Schleswig-Holstein
- Hungary (4):
  - Pécsi Tudományegyetem Klinikai Központ-Bőr-, Nemikórtani és Onkodermatológiai Klinika ( Site 2100), Pécs, Baranya
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Közpo-Department of Dermatology and Allergol, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont-Bőrgyógyászati Klinika ( Site 2102), Debrecen
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz- Onkoradiologiai Osztaly ( Site 2110), Győr
- Israel (4):
  - Emek Medical Center ( Site 2203), Afula
  - Hadassah Medical Center ( Site 2201), Jerusalem
  - Rabin Medical Center ( Site 2202), Petah Tikva
  - Sheba Medical Center ( Site 2200), Ramat Gan
- Italy (6):
  - Instituto Tumori Giovanni Paolo II ( Site 2301), Bari, Apulia
  - Ospedale San Martino-Oncologia Medica 2 ( Site 2303), Genoa, Liguria
  - Istituto Clinico Humanitas-U.O di Oncologia medica ed Ematologia ( Site 2304), Rozzano, Milano
  - Azienda Ospedaliero Universitaria Senese ( Site 2302), Siena, Tuscany
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII-UOC Oncologia ( Site 2305), Bergamo
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-s.c. melanoma, immunoterapia oncologica e terapi, Napoli
- Harbour Cancer & Wellness ( Site 3300), Auckland, New Zealand
- Oslo universitetssykehus, Radiumhospitalet ( Site 2400), Oslo, Norway
- Poland (5):
  - Centrum Medyczne HCP ( Site 2505), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 2501), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 2506), Gdansk, Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakl-Klinika Onkologii Klinicznej, Dzial Ch, Kielce, Świętokrzyskie Voivodeship
- Romania (4):
  - Spitalul Universitar de Urgență Elias ( Site 2600), Bucharest, București
  - SC Radiotherapy Center Cluj SRL-Oncologie Medicala ( Site 2602), Florești, Cluj
  - Centrul de Oncologie Sfantul Nectarie-Medical ( Site 2601), Craiova, Dolj
  - Sigmedical Services SRL ( Site 2603), Suceava
- Spain (8):
  - Hospital Germans Trias i Pujol-Instituto Catalán de Oncología de Badalona ( Site 2804), Badalona, Barcelona
  - HOSPITAL CLÍNIC DE BARCELONA-ICHMO- Clinic Institut of Haematological and Oncological diseases ( Sit, Barcelona, Catalonia
  - Centro Oncologico de Galicia ( Site 2806), A Coruña, Galicia
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 2801), Madrid, Madrid, Comunidad de
  - H.R.U Malaga - Hospital General ( Site 2805), Málaga, Malaga
  - Hospital General Universitario de Valencia-oncology service ( Site 2802), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 2803), Barcelona
  - Clinica Universidad de Navarra-Medical Oncology ( Site 2807), Madrid
- United Kingdom (4):
  - Addenbrooke's Hospital-Cambridge Cancer Trials Centre ( Site 3103), Cambridge, Cambridgeshire
  - Derriford Hospital-Oncology ( Site 3104), Plymouth, Devon
  - Castle Hill Hospital ( Site 3102), Cottingham, East Riding Of Yorkshire
  - Singleton Hospital-South West Wales Cancer Institute ( Site 3100), Swansea

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26309&tenant=MT_MSD_9011